CLINICAL TRIAL: NCT06316635
Title: Evaluation of Microplastics Presence in Otitis Media With Effusion Material
Brief Title: Microplastics in Otitis Media With Effusion Material
Status: Recruiting | Type: Observational
Sponsor: Kerem Kökoğlu (Other)
Responsible Party: Sponsor-Investigator, Kerem Kökoğlu, Principal Investigator, TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: 2023/209; self-funding (Other: Erciyes University)
Record Dates: First submitted 2024-03-10; First posted 2024-03-18 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Microplastics; Otitis Media With Effusion; Biofilms
Keywords: microplastics; hearing loss; otitis media; biofilm; air pollution
MeSH Terms: conditions — Otitis Media with Effusion; Hearing Loss; Otitis Media

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Days
Biospecimen Retention: Samples Without DNA — effusion of otitis media
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient group: patient group has formed as operated patients because of OME A paracentesis and ventilation tube insertion will be performed them. After paracentesis, effusion otitis media will be trapped and sampled for microplastic analysis.
  Interventions: Procedure: ventilation tube insertion

INTERVENTIONS:
Procedure: ventilation tube insertion — a paracentesis will be done to tympanic membrane. Glu will be aspirated and trapped.

SUMMARY:
Microplastic rate is increasing ib athmosphere. They can be found in lung, kidney, heart, even placenta. Otitis media with effusion (OME) is a clinical condition that is ver common in children. Biofilms are blamed in the pathogenesis of OME. Microplastics can include biofilms. Importance of microplastics for potential pathogens and their toxicity aspects should be enlighted with studies. This study aims to investigate presency of microplastics in middle ear fluid of patients with OME.

DETAILED DESCRIPTION:
This study was planned prospectively. With ethical approvel, patients who were followed by bilateral OME at least for three months or one-sided OME at least for 9 months were enrolled to the study. Patients with craniofacial anomaly, cleft palate, had history of previous ear surgery were excluded. They were operated as paracentesis and ventilation tube implementation (VTI). An informed consent form was obtained from them and their parents.

Operation: Surgical indication was made according to disease duration and/or hearing loss. Patients were operated under general anesthesia. Paracentesis was made from posteroinferior quadrant of tympanic membrane. Glu material was trapped in the suction tube and tranferred to glass tubes immediately (Figure 1). For this, glass syringe and 0.9 % serum physiologic were used. Samples were sent from right and left ear seperately. Microplastics determination was made in Enviromental Engineering Labaratory of Faculty of Engineering.

Microplastics Determination Method: It applied according to Prada et. al report (11). Fragments, except blood clots, were washed with a jet of filtered distilled water inside the laminar flow hood to remove any surface contamination and all samples were weighed inside closed glass flasks to the nearest 0.1 mg (Sartorius, Entris, Germany). A method for preparing biological samples for Nile Red staining, previously developed and tested, was followed [16]: (i) incubation for 24 h at 60 °C (Oasis™ Benchtop IR CO2 Incubator, Caron, OH, USA) in 30 mL of 10% KOH (w/v, ≥85%, Labchem, PA, USA); (ii) at 24 h, the temperature was raised to boiling point and the solution immediately filtered on glass fiber filter membrane (1.2 µm pore, Whatman® GF/C, Little Chalfont, Buckinghamshire, UK) mounted in a vacuum glass filtration system; (iii) 100 mL of boiling filtered distilled water was filtered to remove soaps; (iv) 10 mL of acetone was added to the cup for 10 min; (v) an additional 10 mL of acetone was filtered to remove lipophilic matter; (vi) 0.5-1 mL of 0.01 mg mL-1 of Nile Red (microscopy grade, Sigma-Aldrich, St. Louis, MO, USA) was added to the cup for 5 min; (vii) 50 mL of distilled water was filtered; and (viii) stored in glass Petri dishes kept inside cardboard boxes for a week to dry at room temperature (20 °C).

Contamination Control Measures Strict contamination control measures were conducted in all phases, namely by: (i) wearing cotton lab coats and clean gloves; (ii) working in the laminar flow hood in a clean room, maintained by cleaning with ethanol in paper towels followed by cleaning with a duster that attracts and traps dust particles and paper fibers; (iii) filtering all solutions (1.2 µm pore, Whatman® GF/C); (iv) using glass and metal materials; (v) decontaminating glass materials by submerging them in 10% HNO3 for at least 30 min and rinsing with distilled water; (vi) additionally cleaning glass Petri dishes with a N2 air jet; (vii) burning glass microfiber filter membranes at 450 °C for 3 h; (viii) cleaning the cup of the filtration system between samples by dipping it for 15 s in a solution (first batch: acetone, second batch: 30% HNO3) followed by dipping in distilled water; (ix) keeping sample containers closed as much as possible with glass lids, caps, or aluminum foil; and (x) conducting procedural blanks (solutions without samples exposed to sample preparation procedures) for each batch. Each samples were tested by three times for verification. In addition, microplastics were evaluated in serum psyisologic to prevent contamination.

ELIGIBILITY:
Inclusion Criteria:

* patients who were followed by bilateral OME at least for three months or one-sided OME at least for 9 months were enrolled to the study

Exclusion Criteria:

* Patients with craniofacial anomaly, cleft palate, had history of previous ear surgery were excluded

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any age, patients with bilateral OME at least 3 months or unilateral OME at least 9 months
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Microplastic presence | from March 2024 to April 2024
  They will be commented as yes / no. Microplastics Determination Method: It applied according to Prada et. al report. Fragments, except blood clots, were washed with a jet of filtered distilled water inside the laminar flow hood to remove any surface contamination and all samples were weighed inside closed glass flasks to the nearest 0.1 mg (Sartorius, Entris, Germany). A method for preparing biological samples for Nile Red staining, previously developed and tested, was followed.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet I Şahin, Assoc Prof., Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University Medical School, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kokoglu K, Mihciokur H, Uyanik I, Ozturk D, Yildiz H, Tas OB, Kaplan RA. Microplastic presence in the fluid of otitis media with effusion. Int J Pediatr Otorhinolaryngol. 2025 Sep;196:112501. doi: 10.1016/j.ijporl.2025.112501. Epub 2025 Jul 30. PMID 40753682